CLINICAL TRIAL: NCT07393724
Title: Enhancing Tooth Reduction Skill in Fixed Prosthodontics Using Case-Based Learning Among Dental Students: A Quasi-Experimental Study
Brief Title: Enhancing Tooth Reduction Skill in Fixed Prosthodontics Using Case-Based Learning Among Dental Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Moaz Mohamed (Other)
Collaborators: Tanta University (Other)
Responsible Party: Sponsor-Investigator, Dr. Moaz Mohamed, Principal Investigator, Tanta University
Organization: Tanta University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: R-FP-7-25-3209
Record Dates: First submitted 2026-01-23; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Medical Education

STUDY DESIGN:
Intervention Model Description: Participants were assigned to either an educational intervention group or a control group receiving conventional teaching.
Masking Description: This was an open-label educational study with no masking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional teaching group (Active Comparator): Participants received conventional teaching methods as part of the standard fixed prosthodontics curriculum.
  Interventions: Behavioral: Conventional Teaching
- Case-Based Learning (CBL) group (Experimental): Participants received a case-based learning (CBL) educational intervention in fixed prosthodontics.
  Interventions: Behavioral: Case-Based Learning (CBL)

INTERVENTIONS:
Behavioral: Case-Based Learning (CBL) — A structured case-based learning approach was used to support active learning, clinical reasoning, and application of theoretical knowledge during fixed prosthodontics teaching sessions.
  Arms: Case-Based Learning (CBL) group
Behavioral: Conventional Teaching — Traditional lecture-based teaching delivered as part of the standard fixed prosthodontics curriculum.
  Arms: Conventional teaching group

SUMMARY:
This study aimed to evaluate the effectiveness of CBL compared to traditional lecture-demonstration methods in enhancing the foundational knowledge and practical tooth reduction skills of dental students in fixed prosthodontics. Participants were assigned to an experimental group (n=30) receiving four weekly 90-minute CBL sessions and a control group (n=30) receiving traditional lectures and clinical demonstrations

ELIGIBILITY:
Inclusion Criteria:

* Undergraduate preclinical dental students enrolled in the fixed prosthodontics course.
* Students who agreed to participate and provided informed consent.

Exclusion Criteria:

* Students who had previously received formal training in case-based learning (CBL) methodology.
* Students with more than 25% absence rate in regular prosthodontics classes.
* Students who had previously failed the fixed prosthodontics course.
* Individuals with physical limitations that might affect their performance in practical assessments.

Max Age: 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-08-30 (Actual); Study Completion 2025-12-30 (Actual)

PRIMARY OUTCOMES:
Theoretical knowledge examination score | At the end of the educational intervention (up to 4 weeks)
  Students' theoretical knowledge in teeth preparation in fixed prsothdontics was assessed using scores obtained from a structured written theoretical examination (score range: 0-10), where higher scores indicate better theoretical knowledge. The examination was conducted as part of the course assessment.

CONTACTS AND LOCATIONS:
Overall Officials: moaz MO osama ahmed, PHD, Principal Investigator — Faculty of Dentistry, Tanta University
Locations (1):
- Moaz EltoRKY, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No